CLINICAL TRIAL: NCT04827433
Title: Mode of Delivery in Women With Low-lying Placenta: an Italian Multicentre Study
Brief Title: Mode of Delivery in Women With Low-lying Placenta
Acronym: MODEL-PLACENTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: MODEL-PLACENTA STUDY
Record Dates: First submitted 2021-03-22; First posted 2021-04-01 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Low-Lying; Placenta, Hemorrhage, Complicating Delivery
Keywords: low-lying placenta; mode of birth; labor and birth
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women having a persistent low-lying placenta with an IOD between 6 and 20 mm: Women having a persistent low-lying placenta with an IOD between 6 and 20 mm who will be offered a vaginal birth, considering 3 subgroups: 1) 6-10 mm; 2) 11-20mm; 3) > 20 mm (resolution of previa or low-lying placenta)
- Women with normal located placenta: Women with a normally located placenta at the II trimester scan will represent the control group.

SUMMARY:
Multicentre study; observational, longitudinal prospective, case-control

DETAILED DESCRIPTION:
This is a new protocol to evaluate the mode of birth in women with a low-lying placenta. In particular, we intend to propose a vaginal birth in women having a low-lying placenta with a distance between the inferior placental edge and the internal cervical os, called internal-os-distance (IOD) of > 5 mm, as assessed in the late III trimester using transvaginal sonography.

Duration of the study:

* Duration of the study: 54 months
* Duration of enrollment: 42 months
* Duration of follow-up completion of enrolled cases: 6 months
* Duration of data analysis: 6 months

Study Design:

During the II trimester scan, all women presenting a placenta located in the lower uterine segment will undergo evaluation by Transvaginal Sonography (TVS).

If a placenta previa or a low-lying placenta will be confirmed, the woman will be recruited and asked to participate in our study, by signing a written informed consent. In addition women attending the Maternity Triage with vaginal bleeding at < 316/7 weeks of gestation, with a diagnosis of placenta previa or low-lying placenta and not requiring an emergency delivery will be asked to participate and will be recruited after signing the informed consent.

An expert Obstetrician will perform the TVS as scheduled, after inviting the woman to void.

The assessment will include:

* the measurement of the IOD (first caliper on the internal cervical os and second caliper on the inferior placental edge). In case of a marginal sinus, the distance between the internal cervical os and the marginal sinus will also be assessed;
* the cervical length (defined as shortened if ≤25 mm);
* the placental edge thickness, measured within 1 cm from the meeting point between the basal and the chorionic plate. The placental edge will be considered "thick" if > 1cm or if the angle is >45°.

All women with a resolution of a previa or low-lying placenta will be assessed in accordance with the protocol of each participating Maternity Unit, including a scan assessment at 38-39 weeks of gestation or within 28 days from the due date.

Calculation of sample size / power:

Considering that the incidence of previa and low-lying placenta is approximately 2% at the II trimester scan and 0.4% at birth, and assuming a C.I. of 19% in the probability of vaginal birth in women with low-lying placenta/resolved low-lying (> 20 mm), 27 women will be needed for each participating Maternity Unit at the late III trimester scan. Anticipating a 10% drop out, 30 women will be needed to achieve a 95% statistical power to identify a clinically relevant difference in the rate of vaginal birth. This leads to the need of recruiting 150 women at the II trimester scan.

CRF and data management:

All data will be recorded through CRF provided by the promoter center and the database will be based on Microsoft Excel.

A sample of about 20-30 patients for each enrollment center is necessary to have a statistical power of 95% in detecting a clinically relevant difference in outcomes in the various study groups.

Analysis plan:

Descriptive statistics will be performed for all variables evaluated in the study population. Variables will be described by mean and standard deviation if normally distributed, otherwise by median and interquantile range; proportions will be used for categorical variables. The quantitative variables, among the study groups defined by the IOD at the last TVS, will be compared by parametric and non-parametric tests, whereas the categorical variables will be compared using Pearson's chi2 test (Fisher exact test where appropriate). The analyses for the primary outcome measure will be performed among women admitted to labor. A multivariate analysis will be conducted to assess the association between obstetric variables and vaginal birth.

A p-value<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18
* Women with placenta previa or low-lying placenta confirmed by TVS at 19-23 6/7 weeks of gestation.

Women attending Maternity Triage with vaginal bleeding at < 32 weeks of gestation, with a diagnosis of placenta previa or low-lying placenta and not requiring an emergency delivery.

* Women with a normally located placenta at the II trimester ultrasound scan, at 19-23 6/7 week of gestation (control group)
* Single pregnancy
* Signature of the informed consent to participate in the study

Note: Women of the "control group" will be recruited in a 1:3 ratio. After the inclusion of 1 case, 3 women with a normally located placenta will be recruited, according to the parity of the woman representing the case (e.g.: 1 CASE= nulliparous woman, 3 CONTROLS= 3 nulliparous women).

Exclusion Criteria:

* Suspected or confirmed invasive placentation (i.e., placenta accreta)
* Vaginal bleeding requiring emergency delivery
* Inability to meet the conditions set out in the study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women having a persisten low-lying placenta with an IOD between 6 and 20 mm and women with a resolved previa or low-lying placenta with an IOD > 20 mm who will be offered a trial of labor.
  A control group will be represented by women with a normal placental location at the II trimester scan.
Sampling Method: Probability Sample
Enrollment: 2550 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2024-10-28 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of vaginal delivery and urgent cesarean section | Until the end of the study (approximately 54 months).
  Rate of vaginal birth and emergency cesarean section in labor due to vaginal bleeding

SECONDARY OUTCOMES:
Frequency of resolution of placenta previa or low-lying | Until the end of the study (approximately 54 months).
  Frequency of resolution of placenta previa or low-lying in relation to the placental location at the time of diagnosis and in relation to maternal history of hysterotomy
Placental migration speed and its correlation with different variables | Until the end of the study (approximately 54 months).
  Description of time needed for resolution of previa or low-lying placenta in relation to placental location at diagnosis (anterior/posterior; praevia/low-lying), and maternal history of hysterotomy, and its correlation to the mode of birth and risk of bleeding during pregnancy and in labor.
Frequency of ultrasound visualization of the marginal breast in low-lying placentas and other variables | Until the end of the study (approximately 54 months).
  Frequency of marginal sinus in women with low-lying placenta and its relation with mode of birth and risk of ante-, intra-, and post-partum bleeding.
Refusal of elective caesarean section | Until the end of the study (approximately 54 months).
  Rate of women declining the mode of birth suggested by clinicians during counselling.
Morbidity associated with the various groups of placental distance analyzed by the antepartum hemorrhage incidence. | Until the end of the study (approximately 54 months).
  Incidence of antepartum hemorrhage requiring hospital admission or immediate delivery.
Morbidity associated with the various groups of placental distance studied with the intrapartum hemorrhage incidence. | Until the end of the study (approximately 54 months).
  Incidence of intrapartum hemorrhage requiring emergency CS.
Morbidity associated with the various groups of placental distance through the severe postpartum hemorrhage incidence. | Until the end of the study (approximately 54 months).
  Incidence of severe postpartum hemorrhage, defined as bleeding ≥ 1000 ml following birth and administration of uterotonic drugs, use of balloon tamponade, uterine artery embolization, ligature of uterine arteries, hysterectomy, blood transfusion;
Morbidity associated with the various groups of placental distance associated with the admission to Intensive Care Unit (ICU) | Until the end of the study (approximately 54 months).
  The maternal admission to ICU.
Morbidity associated with the various groups of placental distance described by the preterm bith incidence | Until the end of the study (approximately 54 months).
  Incidence of preterm birth can described the morbidity associated wiith the various groups of placenta distance.
Morbidity associated with the various groups of placental distance described through the preterm incidence less than 32 weeks. | Until the end of the study (approximately 54 months).
  Incidence of preterm birth < 32 weeks.
Morbidity associated with the various groups of placental distance according to the neonatal admission to ICU | Until the end of the study (approximately 54 months).
  Neonatal admission to Neonatal ICU and length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ornaghi, Principal Investigator — sara.ornaghi@unimib.it; Patrizia Vergani, Study Director — patrizia.vergani@unimib.it
Locations (17):
- Italy (17):
  - Ospedale Papa Giovanni XXIII, Bergamo
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Ospedale Spedali Civili, Brescia
  - Ospedale Vittorio Emanuele III, Carate Brianza
  - Ospedale M. Bufalini di Cesena, Cesena
  - Ospedale Desio, Desio
  - Ospedale Alessandro Manzoni, Lecco
  - Ospedale dei Bambini "Vittore Buzzi", Milan
  - Ospedale Mangiagalli, Milan
  - Ospedale Niguarda, Milan
  - Ospedale San Raffaele, Milan
  - Ospedale Macedonio Melloni, Milan
  - Ospedale San Paolo, Milan
  - Policlinico di Modena, Modena
  - Obstetrics and Gynecology, MBBM Foundation at San Gerardo Hospital, Monza
  - Ospedale Infermi di Rimini, Rimini
  - Ospedale Filippo Del Ponte, Varese

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Committee on Obstetric Practice. Committee Opinion No. 713: Antenatal Corticosteroid Therapy for Fetal Maturation. Obstet Gynecol. 2017 Aug;130(2):e102-e109. doi: 10.1097/AOG.0000000000002237. PMID 28742678
- [Background] ACOG Committee Opinion No. 764: Medically Indicated Late-Preterm and Early-Term Deliveries. Obstet Gynecol. 2019 Feb;133(2):e151-e155. doi: 10.1097/AOG.0000000000003083. PMID 30681545
- [Background] Al Wadi K, Schneider C, Burym C, Reid G, Hunt J, Menticoglou S. Evaluating the safety of labour in women with a placental edge 11 to 20 mm from the internal cervical Os. J Obstet Gynaecol Can. 2014 Aug;36(8):674-677. doi: 10.1016/S1701-2163(15)30508-9. PMID 25222161
- [Background] Blackwell SC. Timing of delivery for women with stable placenta previa. Semin Perinatol. 2011 Oct;35(5):249-51. doi: 10.1053/j.semperi.2011.05.004. PMID 21962622
- [Background] Bhide A, Prefumo F, Moore J, Hollis B, Thilaganathan B. Placental edge to internal os distance in the late third trimester and mode of delivery in placenta praevia. BJOG. 2003 Sep;110(9):860-4. PMID 14511970
- [Background] Alouini S, Megier P, Fauconnier A, Huchon C, Fievet A, Ramos A, Megier C, Valery A. Diagnosis and management of placenta previa and low placental implantation. J Matern Fetal Neonatal Med. 2020 Oct;33(19):3221-3226. doi: 10.1080/14767058.2019.1570118. Epub 2019 Jan 27. PMID 30688129
- [Background] Dashe JS. Toward consistent terminology of placental location. Semin Perinatol. 2013 Oct;37(5):375-9. doi: 10.1053/j.semperi.2013.06.017. PMID 24176163
- [Background] Farine D, Fox HE, Jakobson S, Timor-Tritsch IE. Vaginal ultrasound for diagnosis of placenta previa. Am J Obstet Gynecol. 1988 Sep;159(3):566-9. doi: 10.1016/s0002-9378(88)80009-7. PMID 3048096
- [Background] Bronsteen R, Valice R, Lee W, Blackwell S, Balasubramaniam M, Comstock C. Effect of a low-lying placenta on delivery outcome. Ultrasound Obstet Gynecol. 2009 Feb;33(2):204-8. doi: 10.1002/uog.6304. PMID 19173234
- [Background] Ginsberg Y, Goldstein I, Lowenstein L, Weiner Z. Measurements of the lower uterine segment during gestation. J Clin Ultrasound. 2013 May;41(4):214-7. doi: 10.1002/jcu.22023. Epub 2013 Mar 16. PMID 23505018
- [Background] Fukuda M, Fukuda K, Shimizu T, Bujold E. Ultrasound Assessment of Lower Uterine Segment Thickness During Pregnancy, Labour, and the Postpartum Period. J Obstet Gynaecol Can. 2016 Feb;38(2):134-40. doi: 10.1016/j.jogc.2015.12.009. Epub 2016 Mar 2. PMID 27032737
- [Background] Jansen C, de Mooij YM, Blomaard CM, Derks JB, van Leeuwen E, Limpens J, Schuit E, Mol BW, Pajkrt E. Vaginal delivery in women with a low-lying placenta: a systematic review and meta-analysis. BJOG. 2019 Aug;126(9):1118-1126. doi: 10.1111/1471-0528.15622. Epub 2019 Mar 10. PMID 30663270
- [Background] Nakamura M, Hasegawa J, Matsuaka R, Mimura T, Ichizuka K, Sekizawa A, Okai T. Amount of hemorrhage during vaginal delivery correlates with length from placental edge to external os in cases with low-lying placenta whose length between placental edge and internal os was 1-2 cm. J Obstet Gynaecol Res. 2012 Aug;38(8):1041-5. doi: 10.1111/j.1447-0756.2011.01776.x. Epub 2012 May 21. PMID 22612540
- [Background] Ohira S, Kikuchi N, Kobara H, Osada R, Ashida T, Kanai M, Shiozawa T. Predicting the route of delivery in women with low-lying placenta using transvaginal ultrasonography: significance of placental migration and marginal sinus. Gynecol Obstet Invest. 2012;73(3):217-22. doi: 10.1159/000333309. Epub 2012 Mar 1. PMID 22378482
- [Background] Jauniaux E, Alfirevic Z, Bhide AG, Belfort MA, Burton GJ, Collins SL, Dornan S, Jurkovic D, Kayem G, Kingdom J, Silver R, Sentilhes L; Royal College of Obstetricians and Gynaecologists. Placenta Praevia and Placenta Accreta: Diagnosis and Management: Green-top Guideline No. 27a. BJOG. 2019 Jan;126(1):e1-e48. doi: 10.1111/1471-0528.15306. Epub 2018 Sep 27. No abstract available. PMID 30260097
- [Background] Oppenheimer L, Holmes P, Simpson N, Dabrowski A. Diagnosis of low-lying placenta: can migration in the third trimester predict outcome? Ultrasound Obstet Gynecol. 2001 Aug;18(2):100-2. doi: 10.1046/j.1469-0705.2001.00450.x. PMID 11529986
- [Background] Oppenheimer L; MATERNAL FETAL MEDICINE COMMITTEE. RETIRED: Diagnosis and management of placenta previa. J Obstet Gynaecol Can. 2007 Mar;29(3):261-266. doi: 10.1016/S1701-2163(16)32401-X. PMID 17346497
- [Background] Oppenheimer LW, Farine D. A new classification of placenta previa: measuring progress in obstetrics. Am J Obstet Gynecol. 2009 Sep;201(3):227-9. doi: 10.1016/j.ajog.2009.06.010. No abstract available. PMID 19733273
- [Background] Reddy UM, Abuhamad AZ, Levine D, Saade GR; Fetal Imaging Workshop Invited Participants. Fetal imaging: executive summary of a joint Eunice Kennedy Shriver National Institute of Child Health and Human Development, Society for Maternal-Fetal Medicine, American Institute of Ultrasound in Medicine, American College of Obstetricians and Gynecologists, American College of Radiology, Society for Pediatric Radiology, and Society of Radiologists in Ultrasound Fetal Imaging Workshop. J Ultrasound Med. 2014 May;33(5):745-57. doi: 10.7863/ultra.33.5.745. PMID 24764329
- [Background] Silver RM. Abnormal Placentation: Placenta Previa, Vasa Previa, and Placenta Accreta. Obstet Gynecol. 2015 Sep;126(3):654-668. doi: 10.1097/AOG.0000000000001005. PMID 26244528
- [Derived] Ornaghi S, Colciago E, Vaglio Tessitore I, Abbamondi A, Antolini L, Locatelli A, Inversetti A, Pintucci A, Cetin I, Bracco B, Fabbri E, Sala V, Meroni M, Volpe G, Benedetti S, Bulfoni C, Marconi A, Lagrasta F, Paolini CL, Mazza E, Candiani M, Valsecchi L, Smid M, Pasi F, Pozzoni M, Castoldi M, Vignali M, Dal Molin G, Guarano A, Pellegrino A, Callegari C, Betti M, Lazzarin S, Prefumo F, Zanardini C, Parolin V, Catalano A, Barbolini E, Antonazzo P, Pignatti L, Tintoni M, Spelzini F, Martinelli A, Facchinetti F, Chiossi G, Vergani P. Mode of birth in women with low-lying placenta: protocol for a prospective multicentre 1:3 matched case-control study in Italy (the MODEL-PLACENTA study). BMJ Open. 2021 Dec 6;11(12):e052510. doi: 10.1136/bmjopen-2021-052510. PMID 34873004